CLINICAL TRIAL: NCT02614157
Title: Lateral Pelvic Lymph Node Dissection After Neoadjuvant Chemo-radiation for Preoperative Enlarged Lateral Nodes in Advanced Low Rectal Cancer: a Phase III Randomized Controlled Trial
Brief Title: Lateral Lymph Node Dissection After Neoadjuvant Chemo-radiation in Advanced Low Rectal Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The enrollment was too low
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Ziqiang Wang,MD, Professor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: pLNR-201501
Record Dates: First submitted 2015-11-23; First posted 2015-11-25 (Estimated); Last update posted 2021-02-01 (Actual); Status verified 2016-06

CONDITIONS: Rectal Cancer
Keywords: rectal cancer; lateral lymph node dissection; neoadjuvant chemoradiation; total mesorectal excision; surgery; recurrence; metastasis; overall survival
MeSH Terms: conditions — Rectal Neoplasms; Recurrence; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LLND+TME group (Experimental): advanced rectal cancer patients after neoadjuvant chem-radiation with suspicious lateral lymph nodes involvement undergo lateral lymph node dissection and total mesorectal excision(LLND+TME)
  Interventions: Procedure: LLND; Device: labeled line
- TME group (No Intervention): advanced rectal cancer patients after neoadjuvant chem-radiation with suspicious lateral lymph nodes involvement undergo total mesorectal excision (TME)solely, without LLND

INTERVENTIONS:
Procedure: LLND — advanced rectal cancer patients whose lymph nodes are suspiciously enlarged after neoadjuvant chemoradiation will undergo lateral lymph node dissection (LLND) and total mesorectal excision (TME)
  Other Names: Lateral Lymph Node Dissection
  Arms: LLND+TME group
Device: labeled line
  Arms: LLND+TME group

SUMMARY:
Lateral lymph nodes (LLD) metastasis is a major cause of local recurrence for advanced rectal cancer. As for the treatment strategies on LLN metastasis, there are huge controversies on whether lateral pelvic lymph nodes dissection (LLND) after neoadjuvant chemo-radiotherapy (nCRT) between Western and Eastern countries. Retrospective cohort evidences indicate that LLND following total mesorectal excision (TME) will bring benefit from cT3-4 rectal cancer, not regular predictive LLND, which will bring more side effects on the contrary. Existing reports tend to recommend LLND for specific individual with suspicious LLN metastasis. Moreover, there is a blank strict prospective randomized control study on the comparison of LLND+TME and LLND after nCRT. Therefore, our trial will compare the efficacy and safety of the two strategies for mid/low rectal cancer with suspicious LLN metastasis. The risk factors (such as radiologic factors, pathologic factors, and serum protein) to predict local recurrence and overall survival will be further investigated.

DETAILED DESCRIPTION:
Recently, the incidence and mortality of colorectal cancer have increased, leading the second prevalence after lung cancer. Local recurrence of mid/low rectal cancer is not only the poor prognostic factor but also the threat of terrible quality of life. Although universal usage of neoadjuvant chemo-radiotherapy (nCRT) and total mesorectal excision (TME) have decreased local recurrence to 5%-10%, the ratio of local recurrence has occupied almost 30% of total metastasis and recurrence incidences, which limited the therapeutic effect of rectal cancer. Increasing evidences have demonstrated lateral pelvic lymph nodes (LLN) metastasis as one of the prominent causes of local recurrence, accompanied with 10%-25% advanced rectal cancer. Published researches also reminder us preoperative LLN involvement may lead to high local recurrence and poor overall survival.

As for the treatment strategies on LLN metastasis, there are huge controversies on whether lateral pelvic lymph nodes dissection (LLND) or LLND+TME after nCRT:

Eastern countries especially Japan favors LLND following TME with the reasons: 1) the incidence of LLN metastasis reaches as high as 10%-25% and 27% of rectal patients who undergo TME solely (without LLND) will develop into local recurrence. And the predictive pelvic recurrence rate will decrease 50%; corresponding 5-year overall survival will increase 8%-9%. 2) efficacy of LLND equals to resection of "local lymph nodes metastases". A large cohort of 11567 cases from Japan demonstrates resection of iliac lymph nodes metastasis does not show any difference from TME of cTxN2aM0 and resection of obturator and external iliac lymph nodes favors that of liver metastasis. 3) Japanese Guidelines for treatment of colorectal in 2014 also recommends mid/low II/III rectal cancer under peritoneal reflex undergo regular TME+LLND.

On the contrary, western countries favor sole TME after nCRT for LLN metastasis, holding that: 1) rate of lymph nodes metastasis is relatively low and LLN metastasis is regarded as systemic metastasis. 2) LLND experiences longer operative time, higher postoperative complications, and poor quality of life. 3) American NCCN and European ESMO guidelines recommend single TME for rectal cancer, if necessary, LLDN is added when LLN is indeed metastasis.

However, there is a blank strict prospective randomized control study on the comparison of nCRT and LLND. Present existing retrospective cohort mainly focus on all the mid/low advanced cancer, not the specific individual of suspicious LLN metastasis. In fact, the results almost indicate no differences on local recurrence and overall survival, except for less operation time, blood loss, and perioperative complications in LLND. Although the latest researches start to report their preliminary outcomes, the patients sample sizes are small and they achieve varied recurrence and overall survival.

In conclusion, the treatment strategy for colorectal cancer has focused on individual and precision. Massive of retrospective reports have indicated that rectal cancer patients with LLN metastasis will benefit from LLND, however, there is hot controversy on the treatment of whether TME+LLND or TME+nCRT for specific rectal patients with suspicious LLN metastasis. Therefore, our trial will compare the efficacy and safety of the two strategies for mid/low rectal cancer with suspicious LLN metastasis. The risk factors (such as radiologic factors, pathologic factors, and serum protein) to predict local recurrence and overall survival will be further investigated.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed rectal cancer (below the peritoneal reflection) Clinical stage I, II, or III
* No extramesorectal lymph node swelling (shorter diameter is less than 10 mm)
* No invasion to other organ (s)
* PS: 0, 1
* No past history of chemotherapy, pelvic surgery or radiation
* Written informed consent operative criteria:
* Mesorectal excision is performed
* Operative findings:
* Main lesion of the tumor is located at the rectum
* Lower tumor margin is below the peritoneal reflection
* R0 after resection

Exclusion Criteria:

* High rectal cancer
* Multiple cancer patients
* Pregnant patients
* Psychological disorder
* Steroid administration
* Cardiac infarction within six months
* Severe pulmonary emphysema and pulmonary fibrosis
* Doctor's decision for exclusion

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2016-05; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
3-year local recurrence | until local-recurrence (up to 3 years)

SECONDARY OUTCOMES:
overall survival | 3 years
disease free survival | 3 years
Incidence of sexual and urinary dysfunction | 1 year
postoperative complications | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ziqiang Wang, MD,PhD, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital, Chengdu, Sichuan, China

REFERENCES:
- [Background] Baik SH, Kim NK, Lee YC, Kim H, Lee KY, Sohn SK, Cho CH. Prognostic significance of circumferential resection margin following total mesorectal excision and adjuvant chemoradiotherapy in patients with rectal cancer. Ann Surg Oncol. 2007 Feb;14(2):462-9. doi: 10.1245/s10434-006-9171-0. Epub 2006 Nov 10. PMID 17096053
- [Background] Quadros CA, Falcao MF, Carvalho ME, Ladeia PA, Lopes A. Metastases to retroperitoneal or lateral pelvic lymph nodes indicated unfavorable survival and high pelvic recurrence rates in a cohort of 102 patients with low rectal adenocarcinoma. J Surg Oncol. 2012 Nov;106(6):653-8. doi: 10.1002/jso.23144. Epub 2012 Apr 25. PMID 22535617
- [Background] Ueno M, Oya M, Azekura K, Yamaguchi T, Muto T. Incidence and prognostic significance of lateral lymph node metastasis in patients with advanced low rectal cancer. Br J Surg. 2005 Jun;92(6):756-63. doi: 10.1002/bjs.4975. PMID 15838895
- [Background] Yano H, Moran BJ. The incidence of lateral pelvic side-wall nodal involvement in low rectal cancer may be similar in Japan and the West. Br J Surg. 2008 Jan;95(1):33-49. doi: 10.1002/bjs.6061. PMID 18165939
- [Background] Kapiteijn E, Marijnen CA, Nagtegaal ID, Putter H, Steup WH, Wiggers T, Rutten HJ, Pahlman L, Glimelius B, van Krieken JH, Leer JW, van de Velde CJ; Dutch Colorectal Cancer Group. Preoperative radiotherapy combined with total mesorectal excision for resectable rectal cancer. N Engl J Med. 2001 Aug 30;345(9):638-46. doi: 10.1056/NEJMoa010580. PMID 11547717
- [Background] Kusters M, Marijnen CA, van de Velde CJ, Rutten HJ, Lahaye MJ, Kim JH, Beets-Tan RG, Beets GL. Patterns of local recurrence in rectal cancer; a study of the Dutch TME trial. Eur J Surg Oncol. 2010 May;36(5):470-6. doi: 10.1016/j.ejso.2009.11.011. Epub 2010 Jan 21. PMID 20096534
- [Background] Nagawa H, Muto T, Sunouchi K, Higuchi Y, Tsurita G, Watanabe T, Sawada T. Randomized, controlled trial of lateral node dissection vs. nerve-preserving resection in patients with rectal cancer after preoperative radiotherapy. Dis Colon Rectum. 2001 Sep;44(9):1274-80. doi: 10.1007/BF02234784. PMID 11584199
- [Background] Ueno H, Mochizuki H, Hashiguchi Y, Ishiguro M, Miyoshi M, Kajiwara Y, Sato T, Shimazaki H, Hase K. Potential prognostic benefit of lateral pelvic node dissection for rectal cancer located below the peritoneal reflection. Ann Surg. 2007 Jan;245(1):80-7. doi: 10.1097/01.sla.0000225359.72553.8c. PMID 17197969
- [Background] Watanabe T, Tsurita G, Muto T, Sawada T, Sunouchi K, Higuchi Y, Komuro Y, Kanazawa T, Iijima T, Miyaki M, Nagawa H. Extended lymphadenectomy and preoperative radiotherapy for lower rectal cancers. Surgery. 2002 Jul;132(1):27-33. doi: 10.1067/msy.2002.125357. PMID 12110792
- [Background] Yano H, Saito Y, Takeshita E, Miyake O, Ishizuka N. Prediction of lateral pelvic node involvement in low rectal cancer by conventional computed tomography. Br J Surg. 2007 Aug;94(8):1014-9. doi: 10.1002/bjs.5665. PMID 17436337
- [Background] Georgiou P, Tan E, Gouvas N, Antoniou A, Brown G, Nicholls RJ, Tekkis P. Extended lymphadenectomy versus conventional surgery for rectal cancer: a meta-analysis. Lancet Oncol. 2009 Nov;10(11):1053-62. doi: 10.1016/S1470-2045(09)70224-4. Epub 2009 Sep 18. PMID 19767239
- [Background] Kim JC, Takahashi K, Yu CS, Kim HC, Kim TW, Ryu MH, Kim JH, Mori T. Comparative outcome between chemoradiotherapy and lateral pelvic lymph node dissection following total mesorectal excision in rectal cancer. Ann Surg. 2007 Nov;246(5):754-62. doi: 10.1097/SLA.0b013e318070d587. PMID 17968166
- [Background] Suzuki K, Muto T, Sawada T. Prevention of local recurrence by extended lymphadenectomy for rectal cancer. Surg Today. 1995;25(9):795-801. doi: 10.1007/BF00311455. PMID 8555697
- [Background] Sato H, Maeda K, Maruta M, Masumori K, Koide Y. Who can get the beneficial effect from lateral lymph node dissection for Dukes C rectal carcinoma below the peritoneal reflection? Dis Colon Rectum. 2006 Oct;49(10 Suppl):S3-12. doi: 10.1007/s10350-006-0699-7. PMID 17106812
- [Background] Kim TH, Jeong SY, Choi DH, Kim DY, Jung KH, Moon SH, Chang HJ, Lim SB, Choi HS, Park JG. Lateral lymph node metastasis is a major cause of locoregional recurrence in rectal cancer treated with preoperative chemoradiotherapy and curative resection. Ann Surg Oncol. 2008 Mar;15(3):729-37. doi: 10.1245/s10434-007-9696-x. Epub 2007 Dec 5. PMID 18057989
- [Background] Kim MJ, Kim TH, Kim DY, Kim SY, Baek JY, Chang HJ, Park SC, Park JW, Oh JH. Can chemoradiation allow for omission of lateral pelvic node dissection for locally advanced rectal cancer? J Surg Oncol. 2015 Mar 15;111(4):459-64. doi: 10.1002/jso.23852. Epub 2015 Jan 5. PMID 25559888
- [Background] Fujita S, Akasu T, Mizusawa J, Saito N, Kinugasa Y, Kanemitsu Y, Ohue M, Fujii S, Shiozawa M, Yamaguchi T, Moriya Y; Colorectal Cancer Study Group of Japan Clinical Oncology Group. Postoperative morbidity and mortality after mesorectal excision with and without lateral lymph node dissection for clinical stage II or stage III lower rectal cancer (JCOG0212): results from a multicentre, randomised controlled, non-inferiority trial. Lancet Oncol. 2012 Jun;13(6):616-21. doi: 10.1016/S1470-2045(12)70158-4. Epub 2012 May 15. PMID 22591948
- [Background] Kobayashi H, Mochizuki H, Kato T, Mori T, Kameoka S, Shirouzu K, Sugihara K. Outcomes of surgery alone for lower rectal cancer with and without pelvic sidewall dissection. Dis Colon Rectum. 2009 Apr;52(4):567-76. doi: 10.1007/DCR.0b013e3181a1d994. PMID 19404054
- [Background] Watanabe T, Itabashi M, Shimada Y, Tanaka S, Ito Y, Ajioka Y, Hamaguchi T, Hyodo I, Igarashi M, Ishida H, Ishiguro M, Kanemitsu Y, Kokudo N, Muro K, Ochiai A, Oguchi M, Ohkura Y, Saito Y, Sakai Y, Ueno H, Yoshino T, Fujimori T, Koinuma N, Morita T, Nishimura G, Sakata Y, Takahashi K, Takiuchi H, Tsuruta O, Yamaguchi T, Yoshida M, Yamaguchi N, Kotake K, Sugihara K; Japanese Society for Cancer of the Colon and Rectum. Japanese Society for Cancer of the Colon and Rectum (JSCCR) guidelines 2010 for the treatment of colorectal cancer. Int J Clin Oncol. 2012 Feb;17(1):1-29. doi: 10.1007/s10147-011-0315-2. Epub 2011 Oct 15. PMID 22002491
- [Background] Dharmarajan S, Shuai D, Fajardo AD, Birnbaum EH, Hunt SR, Mutch MG, Fleshman JW, Lin AY. Clinically enlarged lateral pelvic lymph nodes do not influence prognosis after neoadjuvant therapy and TME in stage III rectal cancer. J Gastrointest Surg. 2011 Aug;15(8):1368-74. doi: 10.1007/s11605-011-1533-7. Epub 2011 May 2. PMID 21533959
- [Background] Akiyoshi T, Ueno M, Matsueda K, Konishi T, Fujimoto Y, Nagayama S, Fukunaga Y, Unno T, Kano A, Kuroyanagi H, Oya M, Yamaguchi T, Watanabe T, Muto T. Selective lateral pelvic lymph node dissection in patients with advanced low rectal cancer treated with preoperative chemoradiotherapy based on pretreatment imaging. Ann Surg Oncol. 2014 Jan;21(1):189-96. doi: 10.1245/s10434-013-3216-y. Epub 2013 Aug 21. PMID 23963871
- [Background] Akiyoshi T, Matsueda K, Hiratsuka M, Unno T, Nagata J, Nagasaki T, Konishi T, Fujimoto Y, Nagayama S, Fukunaga Y, Ueno M. Indications for Lateral Pelvic Lymph Node Dissection Based on Magnetic Resonance Imaging Before and After Preoperative Chemoradiotherapy in Patients with Advanced Low-Rectal Cancer. Ann Surg Oncol. 2015 Dec;22 Suppl 3:S614-20. doi: 10.1245/s10434-015-4565-5. Epub 2015 Apr 21. PMID 25896145
- [Derived] Wei M, Wu Q, Fan C, Li Y, Chen X, Zhou Z, Han J, Wang Z. Lateral pelvic lymph node dissection after neoadjuvant chemo-radiation for preoperative enlarged lateral nodes in advanced low rectal cancer: study protocol for a randomized controlled trial. Trials. 2016 Nov 25;17(1):561. doi: 10.1186/s13063-016-1695-4. PMID 27884204